CLINICAL TRIAL: NCT00101647
Title: A Phase II Study of BMS-354825 in Subjects With Accelerated Phase Chronic Myeloid Leukemia Resistant to or Intolerant of Imatinib Mesylate
Brief Title: Study of Dasatinib (BMS-354825) in Patients With Accelerated Phase Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-005; NCT00108693 (obsolete NCT alias)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Results first posted 2010-03-02 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic myelogenous leukemia (CML): Accelerated phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg, twice daily, until disease progression or intolerable toxicity, switch to the roll-over study or study closure
  Other Names: BMS-354825; Sprycel

SUMMARY:
The purpose of this clinical research study is to learn if BMS-354825 will have activity, defined by hematologic response, in subjects who have accelerated phase chronic myeloid leukemia (CML) who are resistant to or intolerant to imatinib mesylate. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Philadelphia chromosome positive (PH+) or the fused gene BCR/ABL positive (BCR/ABL+) accelerated phase chronic myeloid leukemia (CML) whose disease has primary or acquired hematologic resistance to imatinib mesylate or who are intolerant of imatinib mesylate.
* Subjects must have had prior exposure to imatinib. However, imatinib mesylate does not need to be their most recent CML treatment prior to coming on this study.
* Men and women, 18 years of age or older.
* Adequate hepatic function.
* Adequate renal function.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of least 1 month before and at least 3 months after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Subjects who are eligible and willing to undergo transplantation during the screening period.
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subjects to receive protocol therapy.
* Uncontrolled or significant cardiovascular disease.
* Medications that increase bleeding risk.
* Medications that change heart rhythms.
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
* History of significant bleeding disorder unrelated to CML.
* Concurrent incurable malignancy other than CML.
* Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy.
* Prior therapy with dasatinib (BMS-354825).
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (70):
- United States (21):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Anaheim, California
  - Local Institution, Los Angeles, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Jacksonville, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Kansas City, Kansas
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Detroit, Michigan
  - Local Institution, St Louis, Missouri
  - Local Institution, Hackensack, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Australia (5):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Wien
- Belgium (2):
  - Local Institution, B-Leuven
  - Local Institution, Edegem
- Brazil (3):
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Campinas
- Local Institution, Toronto, Ontario, Canada
- Local Institution, Aarhus, Denmark
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Hamburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Ramat Gan, Israel
- Italy (4):
  - Local Institution, Bologna
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Trondheim, Norway
- Local Institution, Lima, Lima Province, Peru
- Local Institution, Quezon City, Philippines
- Local Institution, Singapore, Singapore
- South Korea (3):
  - Local Institution, Jeollanam-Do
  - Local Institution, Kyunggi-Do
  - Local Institution, Seoul
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Bangkok, Thailand
- United Kingdom (2):
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London

REFERENCES:
- [Background] Guilhot F, Apperley J, Kim DW, Bullorsky EO, Baccarani M, Roboz GJ, Amadori S, de Souza CA, Lipton JH, Hochhaus A, Heim D, Larson RA, Branford S, Muller MC, Agarwal P, Gollerkeri A, Talpaz M. Dasatinib induces significant hematologic and cytogenetic responses in patients with imatinib-resistant or -intolerant chronic myeloid leukemia in accelerated phase. Blood. 2007 May 15;109(10):4143-50. doi: 10.1182/blood-2006-09-046839. Epub 2007 Jan 30. PMID 17264298
- [Background] Apperley JF, Cortes JE, Kim DW, Roy L, Roboz GJ, Rosti G, Bullorsky EO, Abruzzese E, Hochhaus A, Heim D, de Souza CA, Larson RA, Lipton JH, Khoury HJ, Kim HJ, Sillaber C, Hughes TP, Erben P, Van Tornout J, Stone RM. Dasatinib in the treatment of chronic myeloid leukemia in accelerated phase after imatinib failure: the START a trial. J Clin Oncol. 2009 Jul 20;27(21):3472-9. doi: 10.1200/JCO.2007.14.3339. Epub 2009 Jun 1. PMID 19487385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 197 participants were enrolled into the study; 23 participants were not treated (3 participants died, 13 participants no longer met study criteria, 3 participants switched into other studies, 2 participants had adverse events, 1 participant excluded for administrative reasons, and 1 participant withdrew consent).
Groups:
- Imatinib-intolerant: Defined as either: i) toxicity that was considered at least possibly related to imatinib ≤ 400 mg/day that led to a discontinuation of imatinib therapy; ii) ability to tolerate only < 400 mg/day imatinib. A subject who tolerated 400 mg/day imatinib, but was intolerant of higher doses, was not considered imatinib-tolerant.
- Imatinib-resistant: Defined as any of the following: i) initial diagnosis of chronic phase of chronic myeloid leukemia (CML) that progressed to accelerated phase while on treatment with imatinib ≥ 400 mg/day (primary or acquired resistance); ii) initial diagnosis of accelerated phase CML and failure to achieve a hematologic response after ≥ 4 weeks (or ≥ 2 weeks for subjects showing rapid disease progression) of imatinib ≥ 600 mg/day; the required prior imatinib dose was 400 to < 600 mg/day if the subject was intolerant to ≥ 600 mg/day (primary resistance); iii) initial diagnosis of accelerated or blast phase CML that progressed to accelerated phase CML following an initial hematologic response to imatinib ≥ 600 mg/day (acquired resistance). The required prior imatinib dose was 400 to < 600 mg/day if the subject was intolerant of ≥ 600 mg/day.
Period: Overall Study
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Started | 13 (Randomized) | 161 (Randomized)
Completed | 13 | 161
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 13 | 161 | 174
Age, Customized [Number; unit: participants]
  21 to 45 years | 2 | 41 | 43
  46 to 65 years | 6 | 87 | 93
  66 to 75 years | 4 | 25 | 29
  >75 years | 1 | 8 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.2) | 54.5 (13.7) | 54.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 69 | 78
  Male | 4 | 92 | 96
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 23 | 24
  Black or African American | 1 | 8 | 9
  White | 11 | 127 | 138
  Other | 0 | 3 | 3
Performance Status - Eastern Cooperative Oncology Group Scale (ECOG) [Number; unit: units on a scale] — ECOG scale is a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale 0-5, with 0=fully active, able to carry on all pre-disease performance without restriction, and 5=death
  units on a scale
    score=0 fully active | 6 | 73 | 79
    score=1 physically strenuous activity restricted | 4 | 67 | 71
    score=2 capable of all selfcare, unable to work | 3 | 21 | 24
    score=3 limited selfcare, bed/chair confined >50% | 0 | 0 | 0
    score=4 completely disabled, bed/chair confined | 0 | 0 | 0
    score=5 dead | 0 | 0 | 0
Functional Assessment of Cancer Therapy-General (FACT-G) [Mean (Standard Deviation); unit: units on a scale] — FACT-G=27 questions in 4 domains: physical, social/family, emotional, & functional well-being (PWB, SWB, EWB, FWB). Total score=0 to 108; higher score=better health-related quality of life. 12 participants in the Imatinib-Intolerant group had baseline measurements; 130 participants in the Imatinib-Resistant group had baseline measurements for Total FACT-G scores; 134 for PWB; 133 for FWB and SWB; 131 for EWB.
  units on a scale
    Total FACT-G | 81.9 (14.4) | 75.3 (18.0) | 75.8 (17.8)
    Physical Well Being | 22.3 (5.2) | 19.0 (7.1) | 19.2 (7.0)
    Social/Family Well-Being | 22.8 (5.1) | 22.7 (4.8) | 22.7 (4.8)
    Emotional Well-Being | 17.7 (4.8) | 16.7 (4.9) | 16.8 (4.9)
    Functional Well-Being | 19.2 (6.9) | 16.9 (6.7) | 17.1 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Major and Overall Hematologic Response (MaHR and OHR)
Description: MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL). OHR=best confirmed response of MaHR or minor hematologic response (MiHR). Confirmed hematologic response=response confirmed ≥4 weeks after first documented event with no concomitant use of anagrelide or hydroxyurea. Maintaining a response=no 2 consecutive records of nonresponse at assessment. Criteria for CHR and NEL specified in Outcome Measure 2 and criteria for MiHR in Outcome Measure 4.
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during treatment; at end of treatment
Population: All treated subjects
Measure: Number; unit: participants
Groups:
- Imatinib-intolerant: Receiving dasatinib 70 mg twice daily (BID)
- Imatinib-resistant: Receiving dasatinib 70 mg BID
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 13 | 161 | 174
participants
  MaHR | 9 | 103 | 112
  OHR | 12 | 127 | 139

2. Secondary Outcome: Percentage of Participants Who Achieved MaHR and Did Not Progress at 12 Months (Based on the Kaplan-Meier Estimate of the Duration of Response)
Description: MaHR=best response of CHR or NEL. CHR=white blood cells ≤institutional upper limit of normal (iULN); absolute neutrophil count (ANC) ≥1000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes in peripheral blood (PB); bone marrow blasts ≤5%; <5% myelocytes+metamyelocytes in PB; PB basophils ≤ iULN; no extramedullary involvement. NEL=WBC ≤iULN; no blasts/promyelocytes in PB; bone marrow blasts ≤5%; <5% myelocytes+metamyelocytes in PB; PB basophils ≤iULN; no extramedullary involvement; at least 1 of: ANC ≥500/mm3 & <1000/mm3; platelets ≥20,000/mm3 & <100,000/mm3.
Time Frame: 12 months
Population: Population comprised of responders only.
Measure: Number; unit: percentage of responders
Groups:
- Imatinib-intolerant; Imatinib-resistant: Receiving dasatinib 70 mg BID
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 9 | 103 | 112
percentage of responders | 85.7 | 78.3 | 79.0

3. Secondary Outcome: Percentage of Participants Who Achieved MaHR and Did Not Progress at 24 Months in the Imatinib-Resistant Group (Based on the Kaplan-Meier Estimate of the Duration of Response)
Description: Percentage of participants in the Imatinib-Resistant Group who achieved MaHR and did not progress at Month 24, based on the Kaplan-Meier estimate of the duration of response. MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL). Criteria for MaHR and NEL are specified in Outcome Measure 2.
Time Frame: 24 months
Population: Population comprised of responders only. NOTE: Projected duration of MaHR at 24 months in the Imatinib-Intolerant group was beyond the maximum observed time for this cohort, and therefore only the Imatinib-Resistant group is presented.
Measure: Number; unit: percentage of responders
Arm/Group | Imatinib-resistant | Total
Number analyzed (Participants) | 161 | 161
percentage of responders | 60.9 | 59.6

4. Secondary Outcome: Percentage of Participants Who Achieved OHR and Did Not Progress at 12 Months and 24 Months
Description: Percentage of participants who achieved OHR and did not progress at specified timepoints, based on the Kaplan-Meier estimate of the duration of response. OHR=best confirmed response of MaHR or MiHR. MaHR criteria in Outcome Measure 2. MiHR= <15% blasts in bone marrow and <15% blasts in peripheral blood (PB); <30% blasts+promyelocytes in bone marrow and <30% blasts+promyelocytes in PB; <20% basophils in PB; no extramedullary disease other than spleen and liver. Confirmed hematologic response= confirmed ≥4 weeks after 1st documented event with no concomitant use of anagrelide or hydroxyurea.
Time Frame: 12 months, 24 months
Population: Population is comprised of responders only
Measure: Number; unit: Percentage of responders
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 12 | 127 | 139
Percentage of responders
  OHR at 12 months | 69.8 | 69.7 | 69.8
  OHR at 24 months | 34.9 | 51.2 | 50.0

5. Secondary Outcome: Median Time in Days From First Dosing Date to Date of MaHR
Description: as for outcome 2
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during treatment; at end of treatment
Population: Population is comprised of responders only
Measure: Median (Full Range); unit: Days
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 9 | 103 | 112
Days | 84 [28 to 148] | 63 [26 to 420] | 65 [26 to 420]

6. Secondary Outcome: Time to OHR
Description: Median time (in months) from first dosing date to date of OHR. OHR=best confirmed response of MaHR or MiHR. Criteria for MaHR specified in Outcome Measure 2. MiHR= <15% blasts in bone marrow and <15% blasts in peripheral blood (PB); <30% blasts+promyelocytes in bone marrow and <30% blasts+promyelocytes in PB; <20% basophils in PB; no extramedullary disease other than spleen and liver. Confirmed hematologic response = response confirmed ≥4 weeks after 1st documented event with no concomitant use of anagrelide or hydroxyurea.
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during treatment; at end of treatment
Population: Population comprised of responders only
Measure: Median (Full Range); unit: days
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 12 | 127 | 139
days | 34 [28 to 92] | 30 [17 to 420] | 30 [17 to 420]

7. Secondary Outcome: Best Cytogenetic Response
Description: Number of participants with complete, partial, minor, minimal, or no cytogenetic response. Determination of cytogenetic response based on the prevalence (percentage) of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase in a bone marrow sample (aspirates/biopsies).
Time Frame: Baseline (within 4 weeks of therapy start); Every month for Cycles 1-3; Every 12 weeks for Cycles 4+; end of treatment
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 13 | 161 | 174
Participants
  Complete (0% Ph+ metaphases) | 5 | 53 | 58
  Partial (>0% to 35% Ph+ metaphases) | 0 | 12 | 12
  Minor (>35% to 65% Ph+ metaphases) | 0 | 8 | 8
  Minimal (>65% to 95% Ph+ metaphases) | 3 | 37 | 40
  No Response (>95% to 100% Ph+ metaphases) | 4 | 37 | 41
  Unable to determine | 1 | 14 | 15

8. Secondary Outcome: Best Confirmed Hematologic Response
Description: Number of participants with confirmed complete hematologic response (CHR) or No Evidence of Leukemia (NEL), minor hematologic response (MiHR), or no hematologic response. Confirmed hematologic response=response that is confirmed after at least 4 weeks with no concomitant use of anagrelide or hydroxyurea use during this interval. Criteria for CHR and NEL are specified in Outcome Measure 2; criteria for MiHR are specified in Outcome Measure 4.
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during treatment; at end of treatment
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 13 | 161 | 174
Participants
  Complete HR (CHR) | 7 | 80 | 87
  No Evidence of Leukemia (NEL) | 2 | 23 | 25
  Minor HR (MiHR) | 3 | 24 | 27
  No Response | 1 | 34 | 35

9. Secondary Outcome: Number of Participants Who Achieved a Major Molecular Response (MMR) During Treatment Period
Description: Number of participants who achieved an MMR at any time during the treatment period. MMR was calculated by measuring BCR-ABL transcripts in blood during treatment using quantitative reverse transcription-polymerase chain reaction (RT-PCR). BCR-ABL=the fused gene found in subjects with this type of Chronic Myeloid Leukemia (CML).
Time Frame: Baseline, every 12 weeks throughout study (treatment continued until discontinuation due to toxicity, disease progression, or other protocol-specified criteria).
Population: Number of Participants Analyzed=all treated subjects who were assessed for major molecular response; n=participants with or without CCyR in cohort.
Measure: Number; unit: participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 4 | 90 | 94
participants
  MMR in Assessed Participants w/CCyR(n=2;n=39;n=41) | 2 | 17 | 19
  MMR in Assessed Subjects w/o CCyR(n=2;n=51;n=53) | 0 | 11 | 1

10. Secondary Outcome: MaHR and MCyR Among Participants With Baseline BCR-ABL Point Mutations
Description: Major hematologic and cytogenetic responses (MaHR and MCyR) to dasatinib in subjects with mutations at baseline, including imatinib-resistant mutations (IRM) and specific BCR-ABL mutations (SBAM). BCR-ABL=the fused gene found in subjects with this type of CML. Criteria for MaHR are specified in Outcome Measure 2. MCyR=combined complete cytogenetic and partial cytogenetic response rate. Complete Cytogenetic Response= 0% Ph+ Cells in Metaphase in Bone Marrow, Partial Cytogenetic Response > 0% to 35% Ph+ Cells in Metaphase in Bone Marrow.
Time Frame: Baseline, at time of disease progression. (treatment continued until discontinuation due to toxicity, disease progression, or other protocol-specified criteria).
Population: All subjects with baseline mutation data; n=the number of participants with the specified mutation. Baseline mutation data were reported for 162 of the 174 subjects (12/13 imatinib-intolerant and 150/161 imatinib-resistant). At baseline, 89 (59%) imatinib-resistant subjects and 1 imatinib-intolerant subject expressed imatinib resistant mutations.
Measure: Number; unit: Percentage of participants
Groups:
- Participants Achieving MaHR: Percentage of participants achieving MaHR, defined as best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL)
- Participants Achieving MCyR: Percentage of participants achieving major cytogenetic response (MCyR), defined as the rate of complete cytogenetic response (CCyR) plus the rate of partial cytogenetic response (PCyR).
Arm/Group | Participants Achieving MaHR | Participants Achieving MCyR
Number analyzed (Participants) | 162 | 162
Percentage of participants
  Participants with IRM (n=90) | 73 | 40
  with ≥1 IRM in P-loop (n=35) | 69 | 31
  with ≥1 IRM in activation loop (n=15) | 73 | 53
  with ≥1 IRM in P-loop & activation loop (n=3) | 33 | 67
  with ≥1 IRM in other location only (n=43) | 74 | 44
  w/ ≥1 IRM w/2-4-fold increase in IR (n=15) | 87 | 33
  w/ ≥1 IMR w/≥5-fold increase in IR (n=60) | 67 | 35
  SBAM [M244V] at baseline (n=7) | 86 | 71
  SBAM [L248V] at baseline (n=3) | 100 | 67
  SBAM [G250E] at baseline (n=10) | 60 | 20
  SBAM [Y253F/H] at baseline (n=11) | 82 | 45
  SBAM [E255K/V] at baseline (n=11) | 64 | 18
  SBAM [T315I] at baseline (n=9) | 0 | 0
  SBAM [F317L] at baseline (n=4) | 100 | 0
  SBAM [M351T/V] at baseline (n=13) | 85 | 38
  SBAM [E355G] at baseline (n=4) | 50 | 50
  SBAM [F359C/I/V] at baseline (n=12) | 83 | 42
  SBAM [V379I] at baseline (n=6) | 67 | 67
  SBAM [H396R] at baseline (n=6) | 67 | 33
  SBAM [S417Y] at baseline (n=3) | 33 | 0
  SBAM [E459K] at baseline (n=3) | 33 | 100

11. Secondary Outcome: Minimal Clinically Significant Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Number of subjects with minimally significant changes from baseline in the health-related quality of life questionnaire FACT-G. FACT-G=27 questions in 4 domains: physical, social/family, emotional, and functional well-being (PWB, SWB, EWB, FWB). Total score=0 to 108; higher score=better health-related quality of life. Total Score change of 7 or more=minimal clinical important change; PWB, EWB, and FWB score change of 3 or more, and SWB score change of 2 or more=minimal clinically important change.
Time Frame: Baseline, every 2 weeks for the first 3 cycles, following every 4-week cycle, and once at follow-up.(treatment continued until discontinuation due to toxicity, disease progression, or other protocol-specified criteria).
Population: Number of participants with FACT-G assessments at baseline and at least one assessment during treatment
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 12 | 134 | 146
Participants
  Total FACT-G | 5 | 76 | 81
  Physical Well-Being | 4 | 85 | 89
  Social/Family Well-Being | 6 | 50 | 56
  Emotional Well-Being | 7 | 77 | 84
  Functional Well-Being | 4 | 63 | 67

12. Secondary Outcome: Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, Hematologic Toxicities, and Toxicities Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition regardless of causal relationship with treatment. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: Continuous from pretreatment through each 4-week cycle and at follow-up. (treatment continued until discontinuation due to toxicity, disease progression, or other protocol-specified criteria).
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Number analyzed (Participants) | 13 | 161
Participants
  Any AE | 13 | 160
  Grade 3/4 AEs | 12 | 116
  Drug-Related AEs | 13 | 155
  Drug-Related Grade 3-4 AEs | 11 | 95
  Death within 30 days of last dose | 2 | 15
  SAEs | 12 | 113
  Fluid-Retention AEs -Overall | 10 | 104
  Fluid-Retention AEs - Superficial Edema | 8 | 73
  Fluid-Retention AEs -Pleural Effusion | 4 | 60
  Fluid-Retention AEs - Other | 4 | 43
  Grade 3/4 Hematologic Toxicity - Anemia | 11 | 111
  Grade 3/4 Hematologic Toxicity - Thrombocytopenia | 10 | 132
  Grade 3/4 Hematologic Toxicity - Neutropenia | 13 | 120
  Grade 3/4 Hematologic Toxicity - Leukopenia | 11 | 91
  Discontinuations due to Study Drug Toxicity | 2 | 19

13. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib and Its Metabolite BMS-582691 - Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax was obtained from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria,which is also referred to as adjusted R-squared.
Time Frame: Collected on Days 1 and 8 at times as close as possible to the following time points (relative to drug administration): pre-dose, and following drug administration at 30 minutes, 1 hour, 1.5, 2, 3, 4, 5, 6, 8 and 10 hours.
Population: 29 participants had dense PK sampling on Day 1 and Day 8; parameters for 2 participants on Day 8 were excluded due to unreliable data. Participants with all concentration-time values < than the limit of quantitation were treated as missing for PK analysis. n= participants included in the statistical analyses of PK on Day 1 and Day 8, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 29 | 27
ng/mL
  Dasatinib (n=29; n=27) | 69.31 (43.08) | 89.18 (68.38)
  BMS-582691 (n=24; n=24) | 2.81 (1.53) | 4.52 (3.04)

14. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib and Its Metabolite BMS-582691 - Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Time Point Within the Dosing Interval of 12 Hours (AUC[0-T])
Description: The AUC(0-T) was calculated using the mixed log-linear trapezoidal algorithm in Kinetica™. In the calculation of AUC(0-T), predose concentrations that were less than the lower limit of quantitation (LLQ) were assigned a value of zero.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | Day 1 | Day 8
Number analyzed (Participants) | 29 | 27
ng∙h/mL
  Dasatinib (n=29; n=27) | 207.76 (126.05) | 265.02 (184.73)
  BMS-582691 (n=24; n=24) | 9.51 (8.11) | 18.67 (15.58)

15. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib and Its Metabolite BMS-582691 - Time to Maximum Observed Plasma Concentration (Tmax)
Description: The Tmax was obtained from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria,which is also referred to as adjusted R-squared.
Time Frame: as for outcome 13
Population: A total of 29 participants had dense PK sampling on both Day 1 and Day 8; parameters for 2 participants on Day 8 were excluded due to unreliable concentration-time profiles. n=the number of participants on Day 1 and Day 8 who were included in the statistical analyses of PK parameters.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Day 1 | Day 8
Number analyzed (Participants) | 29 | 27
hours
  Dasatinib (n=29; n=27) | 1.26 (0.98) [0.42 to 5.00] | 1.13 (0.93) [0.50 to 4.75]
  BMS-582691 (n=24; n=24) | 1.86 (0.88) [0.50 to 4.32] | 1.75 (1.12) [0.25 to 5.57]

16. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib and Its Metabolite BMS-582691 - Plasma Half-life (T-HALF)
Description: The T-HALF was calculated as Ln2/Lz,where Lz was the absolute value of the slope of the terminal log-linear phase.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Day 1 | Day 8
Number analyzed (Participants) | 29 | 27
hours
  Dasatinib (n=28; n=26) | 3.15 (0.86) | 5.18 (2.12)
  BMS-582691 (n=22; n=20) | 3.30 (1.94) | 5.70 (4.89)

17. Secondary Outcome: Population PK of Dasatinib
Description: Population pharmacokinetic analysis was not done because it is not meaningful for this single study
Time Frame: Day 8 immediately prior to the first daily dose and between 30 minutes to 3 hours following this dose.
Measure: Number; unit: Population PK analysis
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: 160 AEs were reported in Outcome Measure 12. 158 AEs were reported at the 5% threshold.
Arm/Group | Intolerant | Resistant
Serious Adverse Events (participants affected / at risk) | 12/13 | 113/161
Other Adverse Events (participants affected / at risk) | 13/13 | 158/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intolerant (N=13) | Resistant (N=161)
SCLERAL HAEMORRHAGE (Eye disorders) | 0 | 1
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 0
TROPONIN T (Investigations) | 0 | 1
HAEMOGLOBIN (Investigations) | 0 | 1
PLATELET COUNT (Investigations) | 1 | 2
WEIGHT DECREASED (Investigations) | 0 | 1
TROPONIN INCREASED (Investigations) | 1 | 0
TROPONIN T INCREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
BLOOD CULTURE POSITIVE (Investigations) | 0 | 1
FIBRIN D DIMER INCREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1
GRANULOCYTE COUNT DECREASED (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 1
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 0 | 1
PALPITATIONS (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 0 | 1
COR PULMONALE (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
CARDIAC DISORDER (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
FLUSHING (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 2
HAEMORRHAGE (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 0 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0
THYROIDITIS (Endocrine disorders) | 1 | 0
MANIA (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 3
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1
AUTOIMMUNE DISORDER (Immune system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
FACIAL PALSY (Nervous system disorders) | 0 | 1
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 | 1
MENINGEAL DISORDER (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 4
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 2
COLITIS (Gastrointestinal disorders) | 1 | 1
MELAENA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 4
DIARRHOEA (Gastrointestinal disorders) | 1 | 9
GASTRITIS (Gastrointestinal disorders) | 0 | 1
PROCTITIS (Gastrointestinal disorders) | 0 | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 2
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 2
PERIODONTITIS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 4
ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 11
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 3
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 0 | 1
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 5
CHOLERA (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 1 | 4
PNEUMONIA (Infections and infestations) | 2 | 15
SINUSITIS (Infections and infestations) | 0 | 1
VARICELLA (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 1
ERYSIPELAS (Infections and infestations) | 0 | 2
SEPTIC SHOCK (Infections and infestations) | 1 | 2
HERPES ZOSTER (Infections and infestations) | 0 | 2
ANAL INFECTION (Infections and infestations) | 0 | 1
OTITIS EXTERNA (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
MENINGITIS VIRAL (Infections and infestations) | 0 | 1
PERIANAL ABSCESS (Infections and infestations) | 0 | 1
PULMONARY MYCOSIS (Infections and infestations) | 0 | 1
SALMONELLA SEPSIS (Infections and infestations) | 0 | 1
INFECTIVE MYOSITIS (Infections and infestations) | 0 | 1
SEPSIS PASTEURELLA (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 1
INFECTED SEBACEOUS CYST (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 0 | 3
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 2
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
SPLENECTOMY (Surgical and medical procedures) | 0 | 1
BONE MARROW TRANSPLANT (Surgical and medical procedures) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 2 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 15
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 13
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
GRANULOMA ANNULARE (Skin and subcutaneous tissue disorders) | 0 | 1
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 1
OEDEMA GENITAL (Reproductive system and breast disorders) | 0 | 1
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 10
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 5
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 31
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 4
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 8
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHILLS (General disorders) | 0 | 1
OEDEMA (General disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 2
PYREXIA (General disorders) | 1 | 21
ASTHENIA (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 0 | 1
ADVERSE EVENT (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 2
INFUSION RELATED REACTION (General disorders) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
TUMOUR LYSIS SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 10
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intolerant (N=13) | Resistant (N=161)
EYE SWELLING (Eye disorders) | 1 | 2
VISION BLURRED (Eye disorders) | 1 | 8
VITREOUS FLOATERS (Eye disorders) | 1 | 1
SCLERAL HAEMORRHAGE (Eye disorders) | 1 | 1
EYELID FUNCTION DISORDER (Eye disorders) | 1 | 0
CARDIAC MURMUR (Investigations) | 1 | 11
PLATELET COUNT (Investigations) | 1 | 6
NEUTROPHIL COUNT (Investigations) | 1 | 1
WEIGHT DECREASED (Investigations) | 1 | 36
WEIGHT INCREASED (Investigations) | 2 | 34
PLATELET COUNT DECREASED (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 9
PALPITATIONS (Cardiac disorders) | 1 | 11
CARDIAC FAILURE (Cardiac disorders) | 1 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 6
PERICARDIAL DISEASE (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 13
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 1 | 0
PALLOR (Vascular disorders) | 1 | 3
FLUSHING (Vascular disorders) | 1 | 12
HAEMATOMA (Vascular disorders) | 1 | 16
HYPOTENSION (Vascular disorders) | 0 | 10
LYMPHOEDEMA (Vascular disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 13
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 1
THYROID PAIN (Endocrine disorders) | 1 | 0
HYPOTHYROIDISM (Endocrine disorders) | 1 | 1
ANXIETY (Psychiatric disorders) | 1 | 11
INSOMNIA (Psychiatric disorders) | 0 | 17
DEPRESSION (Psychiatric disorders) | 4 | 10
LOSS OF LIBIDO (Psychiatric disorders) | 1 | 0
SLEEP DISORDER (Psychiatric disorders) | 1 | 1
LIBIDO DECREASED (Psychiatric disorders) | 1 | 1
HEPATOMEGALY (Hepatobiliary disorders) | 1 | 1
SEASONAL ALLERGY (Immune system disorders) | 1 | 4
TREMOR (Nervous system disorders) | 1 | 5
HEADACHE (Nervous system disorders) | 7 | 77
DIZZINESS (Nervous system disorders) | 4 | 29
DYSGEUSIA (Nervous system disorders) | 1 | 7
PARAESTHESIA (Nervous system disorders) | 1 | 10
HYPOAESTHESIA (Nervous system disorders) | 1 | 5
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 1
NAUSEA (Gastrointestinal disorders) | 5 | 73
ASCITES (Gastrointestinal disorders) | 1 | 2
COLITIS (Gastrointestinal disorders) | 1 | 8
VOMITING (Gastrointestinal disorders) | 7 | 46
DIARRHOEA (Gastrointestinal disorders) | 10 | 106
DRY MOUTH (Gastrointestinal disorders) | 1 | 5
DYSPEPSIA (Gastrointestinal disorders) | 2 | 17
DYSPHAGIA (Gastrointestinal disorders) | 2 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 11
ORAL PAIN (Gastrointestinal disorders) | 2 | 4
TOOTHACHE (Gastrointestinal disorders) | 0 | 12
FLATULENCE (Gastrointestinal disorders) | 1 | 11
STOMATITIS (Gastrointestinal disorders) | 3 | 15
FAECES HARD (Gastrointestinal disorders) | 1 | 0
SIGMOIDITIS (Gastrointestinal disorders) | 1 | 0
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 31
HAEMORRHOIDS (Gastrointestinal disorders) | 3 | 13
MOUTH PLAQUE (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 3 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 46
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 10
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 14
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 10
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 12
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 18
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 19
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 12
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 3
TINNITUS (Ear and labyrinth disorders) | 1 | 2
INFLUENZA (Infections and infestations) | 1 | 12
PNEUMONIA (Infections and infestations) | 2 | 10
SINUSITIS (Infections and infestations) | 0 | 10
BRONCHITIS (Infections and infestations) | 0 | 15
CELLULITIS (Infections and infestations) | 1 | 5
LARYNGITIS (Infections and infestations) | 2 | 3
BACTERAEMIA (Infections and infestations) | 1 | 2
ORAL HERPES (Infections and infestations) | 0 | 13
PHARYNGITIS (Infections and infestations) | 3 | 10
SALMONELLOSIS (Infections and infestations) | 1 | 0
GENITAL HERPES (Infections and infestations) | 1 | 1
LUNG INFECTION (Infections and infestations) | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 25
ORAL CANDIDIASIS (Infections and infestations) | 2 | 5
GENITAL CANDIDIASIS (Infections and infestations) | 1 | 0
CATHETER SITE INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 14
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 25
NOCTURIA (Renal and urinary disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 2 | 39
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 6
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 10
ANAEMIA (Blood and lymphatic system disorders) | 1 | 17
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 12
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 18
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 1
ACNE (Skin and subcutaneous tissue disorders) | 1 | 10
RASH (Skin and subcutaneous tissue disorders) | 6 | 53
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 13
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 13
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 20
PETECHIAE (Skin and subcutaneous tissue disorders) | 2 | 34
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 5
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 6
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 12
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 6
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 4
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 3
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 2 | 9
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 2
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 1 | 1
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 | 2
BREAST ENGORGEMENT (Reproductive system and breast disorders) | 1 | 0
PENILE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 1
EJACULATION DISORDER (Reproductive system and breast disorders) | 1 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 2 | 2
INJURY (Injury, poisoning and procedural complications) | 1 | 0
SUNBURN (Injury, poisoning and procedural complications) | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 11
JOINT SPRAIN (Injury, poisoning and procedural complications) | 1 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 8
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 32
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 34
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 22
NECK MASS (Musculoskeletal and connective tissue disorders) | 1 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 46
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 12
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 2
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 39
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 25
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 5
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 60
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 60
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 25
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 9
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 8
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 52
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 8
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 29
PAIN (General disorders) | 0 | 15
CHILLS (General disorders) | 6 | 23
FATIGUE (General disorders) | 8 | 65
MALAISE (General disorders) | 1 | 4
PYREXIA (General disorders) | 10 | 76
ASTHENIA (General disorders) | 3 | 37
CHEST PAIN (General disorders) | 3 | 14
FACE OEDEMA (General disorders) | 0 | 12
FEELING COLD (General disorders) | 1 | 2
CHEST DISCOMFORT (General disorders) | 2 | 8
OEDEMA PERIPHERAL (General disorders) | 6 | 56
GENERALISED OEDEMA (General disorders) | 2 | 2
MUCOSAL INFLAMMATION (General disorders) | 1 | 9
INFLAMMATION OF WOUND (General disorders) | 1 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 2 | 0
CATHETER SITE RELATED REACTION (General disorders) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.